CLINICAL TRIAL: NCT03556995
Title: Score Scale to Assess Risk of Bleeding in Bariatric Surgery
Brief Title: Suggesting Score Scale for Risk of Bleeding in Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, head of the department of general surgery, Assuta Medical Center
Other Study IDs: 01-18
Record Dates: First submitted 2018-06-03; First posted 2018-06-14 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Bariatric Surgery Candidate; Complication; Bleeding
MeSH Terms: conditions — Obesity; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric surgery patients: All patients above 18 that underwent bariatric surgery
  Interventions: Other: bariatric surgery patients

INTERVENTIONS:
Other: bariatric surgery patients

SUMMARY:
As bleeding is a major risk in bariatric surgeries, we aimed our study to find any predictors to such bleeding within the surgery or 30 days after surgery. The study is a retrospective study collecting patients data, surgeons data, and hospitals data in order to find if any of the factors influencing patients, surgeons or hospitals, has to do with bleeding in these surgeries and if it does impact bleeding in what way. The goal is finding a predictor that it's neutralizing may prevent bleeding in bariatric surgeries.

DETAILED DESCRIPTION:
Were collected retrospectively the data of all patients (age 18 and older) that underwent bariatric surgery in Assuta Hospitals (Assuta is a nationwide privet hospitals network), during the years 2013-2016.

Patients underwent one of three procedures:

* laparoscopic sleeve gastrectomy (LSG),
* laparoscopic gastrectomy by-pass (LGBP)
* laparoscopic adjustable gastric band (LAGB) Demographic data of patients was collected (age, gender. BMI, habits, smoking, alcohol consumption etc.), as well as medical history, background diseases, family medical history, previous surgeries and procedures, chronic treatments, use of medications etc., We have also collected surgeons and hospital data - in which hospital was the surgery done? Surgery technique, surgeon's experience, capacity of surgeon - how many bariatric surgeries are done by the surgeon per months? Statistical analyses was done using chi square and Fisher's exact test for analyzing specific single variables. When analyzing the possible connection between BMI and bleeding, BMI values were split into three categories 30<BMI<35, 35<BMI<40 and BMI>40. The use of single variable analyses enabled us to focus on a relatively small number of variables in the multivariable analyses. Variables that were statistically significant (p<0.05) were used as independent variables in logistic regression tests.

ELIGIBILITY:
Inclusion Criteria:all patients that underwent bariatric surgery -

Exclusion Criteria: Under 18 years old

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that underwent any bariatric surgery in Assuta medical network, composed by 4 hospital of High Volume of bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 9044 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
operative or postoperative bleeding complication | 30 days postoperative
  patients underwent any type of bariatric surgery in our medical network

SECONDARY OUTCOMES:
treatment of the complication | 30 days postoperative
  Treated conservatively, re operation, endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta MC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
No IPD sharing Data

REFERENCES:
- [Result] Buchwald H, Oien DM. Metabolic/bariatric surgery worldwide 2011. Obes Surg. 2013 Apr;23(4):427-36. doi: 10.1007/s11695-012-0864-0. PMID 23338049
- [Result] Sovik TT, Aasheim ET, Taha O, Engstrom M, Fagerland MW, Bjorkman S, Kristinsson J, Birkeland KI, Mala T, Olbers T. Weight loss, cardiovascular risk factors, and quality of life after gastric bypass and duodenal switch: a randomized trial. Ann Intern Med. 2011 Sep 6;155(5):281-91. doi: 10.7326/0003-4819-155-5-201109060-00005. PMID 21893621
- [Result] Adams TD, Davidson LE, Litwin SE, Kolotkin RL, LaMonte MJ, Pendleton RC, Strong MB, Vinik R, Wanner NA, Hopkins PN, Gress RE, Walker JM, Cloward TV, Nuttall RT, Hammoud A, Greenwood JL, Crosby RD, McKinlay R, Simper SC, Smith SC, Hunt SC. Health benefits of gastric bypass surgery after 6 years. JAMA. 2012 Sep 19;308(11):1122-31. doi: 10.1001/2012.jama.11164. PMID 22990271
- [Result] Courcoulas AP, Christian NJ, Belle SH, Berk PD, Flum DR, Garcia L, Horlick M, Kalarchian MA, King WC, Mitchell JE, Patterson EJ, Pender JR, Pomp A, Pories WJ, Thirlby RC, Yanovski SZ, Wolfe BM; Longitudinal Assessment of Bariatric Surgery (LABS) Consortium. Weight change and health outcomes at 3 years after bariatric surgery among individuals with severe obesity. JAMA. 2013 Dec 11;310(22):2416-25. doi: 10.1001/jama.2013.280928. PMID 24189773
- [Result] Suter M, Calmes JM, Paroz A, Giusti V. A 10-year experience with laparoscopic gastric banding for morbid obesity: high long-term complication and failure rates. Obes Surg. 2006 Jul;16(7):829-35. doi: 10.1381/096089206777822359. PMID 16839478
- [Result] Nielsen AW, Helm MC, Kindel T, Higgins R, Lak K, Helmen ZM, Gould JC. Perioperative bleeding and blood transfusion are major risk factors for venous thromboembolism following bariatric surgery. Surg Endosc. 2018 May;32(5):2488-2495. doi: 10.1007/s00464-017-5951-9. Epub 2017 Nov 3. PMID 29101558
- [Result] Fecso AB, Samuel T, Elnahas A, Sockalingam S, Jackson T, Quereshy F, Okrainec A. Clinical Indicators of Postoperative Bleeding in Bariatric Surgery. Surg Laparosc Endosc Percutan Tech. 2018 Feb;28(1):52-55. doi: 10.1097/SLE.0000000000000480. PMID 29023333
- [Result] Daigle CR, Brethauer SA, Tu C, Petrick AT, Morton JM, Schauer PR, Aminian A. Which postoperative complications matter most after bariatric surgery? Prioritizing quality improvement efforts to improve national outcomes. Surg Obes Relat Dis. 2018 May;14(5):652-657. doi: 10.1016/j.soard.2018.01.008. Epub 2018 Jan 12. PMID 29503096
- [Result] Nguyen NT, Paya M, Stevens CM, Mavandadi S, Zainabadi K, Wilson SE. The relationship between hospital volume and outcome in bariatric surgery at academic medical centers. Ann Surg. 2004 Oct;240(4):586-93; discussion 593-4. doi: 10.1097/01.sla.0000140752.74893.24. PMID 15383786
- [Result] Nimeri AA, Bautista J, Ibrahim M, Philip R, Al Shaban T, Maasher A, Altinoz A. Mandatory Risk Assessment Reduces Venous Thromboembolism in Bariatric Surgery Patients. Obes Surg. 2018 Feb;28(2):541-547. doi: 10.1007/s11695-017-2909-x. PMID 28836135
- [Result] Colquitt JL, Pickett K, Loveman E, Frampton GK. Surgery for weight loss in adults. Cochrane Database Syst Rev. 2014 Aug 8;2014(8):CD003641. doi: 10.1002/14651858.CD003641.pub4. PMID 25105982